CLINICAL TRIAL: NCT03663335
Title: A Partially-blinded, Active-controlled, Multicenter, Randomized Study Evaluating Efficacy, Safety, Tolerability, Pharmacokinetic (PK) and Pharmacodynamic (PD) of an Anti-CD40 Monoclonal Antibody, CFZ533, in de Novo and Maintenance Kidney Transplant Recipients (CIRRUS I)
Brief Title: Study of Efficacy, Safety, Tolerability, Pharmacokinetic (PK) and Pharmacodynamic (PD) of an Anti-CD40 Monoclonal Antibody, CFZ533, in Kidney Transplant Recipients
Acronym: CIRRUS I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCFZ533A2201; 2017-003607-22 (EudraCT Number); CCFZ533A2201 (Other: Novartis); 03663335 (Other: Clinicaltrials.gov)
Record Dates: First submitted 2018-06-04; First posted 2018-09-10 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Kidney Transplant Rejection
Keywords: Renal transplantation, CFZ533, CNI-free immunosuppression, transplant rejection, allograft rejection.

STUDY DESIGN:
Intervention Model Description: Study CCFZ533A2201 is a randomized, 60-month, active-controlled, partially-blinded, multicenter, dose range finding study to evaluate the efficacy, safety, tolerability, PK and PD of CFZ533 in 2 different cohorts, as compared to standard of care comprised of tacrolimus, MMF and corticosteroids.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1/Cohort 1 (Experimental): CFZ533 dose A+ MMF + Corticosteroids
  Interventions: Biological: CFZ533 - MMF - CS
- Arm 2/Cohort 1 (Experimental): CFZ533 dose B + MMF + Corticosteroids
  Interventions: Biological: CFZ533 - MMF - CS
- Arm 3/Cohort 1 (Active Comparator): Control/Standard of Care: TAC + MMF + Corticosteroids
  Interventions: Drug: Tacrolimus - MMF - +/- corticosteroids
- Arm 1/Cohort 2 (Experimental): CFZ533 dose C + MMF ± Corticosteroids
  Interventions: Biological: CFZ533 - MMF - CS
- Arm 2/Cohort 2 (Active Comparator): Tac + MMF ± Corticosteroids
  Interventions: Drug: Tacrolimus - MMF - +/- corticosteroids

INTERVENTIONS:
Biological: CFZ533 - MMF - CS — Comparison with standard of care immunosuppression
  Arms: Arm 1/Cohort 1; Arm 1/Cohort 2; Arm 2/Cohort 1
Drug: Tacrolimus - MMF - +/- corticosteroids — Standard of care immunosupprevive regimen
  Arms: Arm 2/Cohort 2; Arm 3/Cohort 1

SUMMARY:
The purpose of this study is to investigate the safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of three CFZ533 dose regimens in kidney transplant recipients.

This study will allow assessment of the ability of CFZ533 to replace Calcineurin inhibitors (CNIs) in terms of anti-rejection efficacy, while providing better renal function with a better safety and tolerability profile. Results of this study will be used to inform the CFZ533 dose and regimen selection for investigation in later phases of clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any assessment.
* Male or female patient ≥ 18 years old.
* Up to date vaccination as per local immunization schedules.
* Recipients of a kidney transplant
* Recipients of a primary kidney transplant from a heart-beating deceased, living unrelated or non-HLA identical living related donors.

Exclusion Criteria:

* Multi-organ transplant recipients or prior kidney transplant.
* Recipients of an organ from a non-heart beating donor.
* Recipient of an organ from an HLA identical living related donor.
* ABO incompatible or complement-dependent lymphocytotoxic (CDC) crossmatch positive transplant
* Recipients of kidneys from donors who are older than 65 years.
* Recipients of kidneys from donors with terminal serum creatinine > 2 mg/dL.
* Patients at high immunological risk for rejection
* Patient who is anti-HIV positive, HBsAg-positive or anti-HCV positive (without proof of sustained viral response (SVR) after anti-HCV treatment).
* Recipient of a kidney from a donor who tests positive for HIV, HBsAg/HBc positive or HCV.
* A negative Epstein Barr virus (EBV) test.
* Evidence of advanced liver disease (Child-Pugh C), or any sign of liver decompensation.
* Patient with severe systemic infections, current or within the two weeks prior to randomization.
* History of malignancy of any organ system, treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases, with the exception of localized excised non-melanomatous skin lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with composite event (BPAR, Graft Loss or Death) | Month 12
  Cohorts 1 and 2-Proportion of patients with composite event (BPAR, Graft Loss or Death) over 12 months

SECONDARY OUTCOMES:
Cohorts 1 and 2-Mean eGFR over 12 months | Baseline to month 12
  Renal function at Month 12
Cohorts 1 and 2-Cohorts 1 and 2-safety of CFZ533 regimens compared to a tacrolimus based regimen | Baseline to month 12
  Proportion of patients with AEs, SAEs, infections, malignancies, thromboembolic events, major adverse cardiovascular events, new onset diabetes mellitus (NODM).
Cohorts 1 and 2-Cohorts 1 and 2 - tolerability of CFZ533 regimens compared to a tacrolimus based regimen | Baseline to month 12
  Tolerability assessment by rate of premature discontinuation from study, premature discontinuation of study drug, dose interruption and dose adjustment
Cohorts 1 and 2-pharmacokinetics of CFZ533 during the 60 months treatment period and explore the dose-exposure relationship | Baseline to month 60
  Free CFZ533 plasma concentrations over time
Cohorts 1 and 2-immunogenicity of CFZ533 during the 60 months treatment period | Baseline to month 60
  Semi-quantitative analysis of anti-CFZ533 antibodies in plasma

CONTACTS AND LOCATIONS:
Locations (68):
- United States (13):
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Seattle, Washington
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
- Australia (3):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Clayton, Victoria
- Novartis Investigative Site, Leuven, Belgium
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Vancouver, British Columbia, Canada
- Novartis Investigative Site, Prague, Czechia
- France (8):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
- Germany (8):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Mainz
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Japan (8):
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Tomigusuku, Okinawa
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Riga, Latvia
- Netherlands (3):
  - Novartis Investigative Site, Utrecht, The Netherlands
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Seoul, South Korea
- Spain (4):
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Zaragoza
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Uppsala
- Novartis Investigative Site, Bern, Switzerland
- United Kingdom (3):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com